# Statistical Analysis Plan (SAP)

# Evaluation of the Precision and Sensitivity of Tilmanocept Uptake Value (TUV) on Tc 99m Tilmanocept Planar Imaging

Study No: NAV3-31

Version 1.1

July 6, 2021

Prepared for Navidea Biopharmaceuticals, Inc. 4995 Bradenton Avenue, Suite 240 Dublin, OH 43017

Prepared by
STATKING Clinical Services
759 Wessel Drive
Fairfield, OH 45014
513-858-2989
www.statkingclinical.com



# **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

I agree to the format and content of this document.

Approved by:

Michael Rosol, PhD Chief Medical Officer Navidea Biopharmaceuticals

4995 Bradenton Avenue, Suite 240

Dublin, Ohio 43017 MRosol@navidea.com Date

Bonnie Abbruzzese, MS, CCRA

Senior Director, Clinical Research & Operations

Navidea Biopharmaceuticals

4995 Bradenton Avenue, Suite 240

Dublin, Ohio 43017

BAbbruzzese@navidea.com

Authored by:

Lori Christman, PhD Director of Biostatistics STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 317 lori@statkingclinical.com 07/07/202/ Date

| Approved I | by ( | (internal | review) | : |
|------------|------|-----------|---------|---|
|------------|------|-----------|---------|---|

lan Lees, MS Statistician

STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 327 ian@statkingclinical.com Date

Approved by:

Clare Geiger, RN Project Manager

**STATKING Clinical Services** 

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 304 clare@statkingclinical.com 7-7-2021

Date

# **Revision History**

#### Version 1.0 to 1.1:

- Updated the TUV prediction algorithms 1 and 4 in Section 4.2.2 to include a 10% decrease as a predicted responder. The prior SAP version defined a responder as one with a strictly greater than 10% decrease.
- Added clarification in Section 4.2.2 that the TUV prediction algorithms are to be implemented after rounding the change in TUV calculations to the nearest integer percentage (i.e., nearest hundredths place for a proportion).

# **List of Abbreviations and Definitions of Terms**

| Term | Definition |
|---|---|
| Δ | Greek letter delta, used to represent the change in a |
| | particular variable |
| μg | microgram |
| ACPA | anti-citrullinated protein/peptide antibody |
| ACR/EULAR | American College of Rheumatology/ European League |
| | Against Rheumatism |
| AE | adverse event |
| Anti-TNF-α | Anti-Tumor Necrosis Factor $\alpha$ biological Disease Modifying |
| bDMARD | Anti-Rheumatic Drug |
| CDAI | Clinical Disease Activity Index |
| CFB | change from baseline |
| CI | confidence interval |
| CRF | case report form |
| CSR | clinical study report |
| CT | X-ray computed tomography |
| CV | coefficient of variation |
| DAS28 | Disease activity score used with the ACR/EULAR 2010 RA |
| | guidelines |
| ECG | electrocardiogram |
| FDA | Food and Drug Administration |
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| HC(s) | healthy control(s) |
| ICH | International Conference on Harmonization |
| ITD | intent-to-diagnose |
| IV | intravenous |
| mCi | milliCurie (37x10 <sup>6</sup> becquerels; 37megabecquerels) |
| MCP | metacarpophalange |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NPV | Negative Predictive Value |
| OA | Osteoarthritis or Overall Accuracy, depending on context |
| PIP | proximal interphalange |
| PP | per protocol |
| PPV | Positive Predictive Value |
| RA | rheumatoid arthritis |
| ROI | region of interest |
| RR | reference region |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SOC | system organ class |
| SPECT | single photon emission computed tomography |

| Term | Definition |
|---|---|
| Tc 99m | technetium-99m metastable isotope; γ-emitting (half-life |
| | 6.02 h) |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| tilmanocept | DTPA Mannosyl Dextran (the US Adopted Name for the |
| | drug substance of Lymphoseek) |
| TUV | Tilmanocept uptake value |
| US | United States |
| $\bar{X}_{BRAIN}$ | the decay-corrected average voxel intensity of the brain |
| | RR of a subject at the anterior view at 1 or 3-hours post- |
| | injection |
| $\bar{X}_{ROI}$ | the decay-corrected average voxel intensity of a region of |
| | interest |

# **Table of Contents**

| APPROVAL PAGE | 1 |
|------------------------------------------------------|----|
| REVISION HISTORY | 4 |
| LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 5 |
| INTRODUCTION | 9 |
| 1.0 SYNOPSIS OF STUDY DESIGN/PROCEDURES | 9 |
| 1.1 Design and Treatment | 10 |
| 1.2 Study Procedures | 10 |
| 1.3 Sample Size | 12 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 13 |
| 2.1 Types of Analyses | 13 |
| 2.2 Analysis Populations | 13 |
| 2.3 Missing Data Conventions | 13 |
| 2.4 Interim Analyses | 13 |
| 2.5 Calculation of TUV | 14 |
| 2.6 Study Center Considerations in the Data Analysis | 16 |
| 2.7 Documentation and Other Considerations | 16 |
| 3.0 ANALYSIS OF BASELINE PATIENT CHARACTERISTICS | 17 |
| 4.0 ANALYSIS OF EFFICACY | 17 |
| 4.1 Description of Efficacy Variables | 17 |
| 4.2 Analysis of Efficacy Variables | 21 |
| 5.0 ANALYSIS OF SAFETY | 27 |
| 5.1 Description of Safety Variables | 27 |

| 5.2 Description of Safety Analysis | 27 |
|---------------------------------------------------------|----|
| 6.0 OTHER RELEVANT DATA ANALYSES/SUMMARIES | 29 |
| 6.1 Patient Completion | 29 |
| 6.3 Study Drug Administration | 29 |
| 6.4 RA Evaluation and Screening Physical Exam | 29 |
| 6.5 Concomitant Medications | 29 |
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 31 |
| 9.0 REFERENCES | 35 |
| APPENDIX A – TABLES, FIGURES AND LISTING SPECIFICATIONS | 36 |
| ADDENINIV D. TARI E CHELL C | 20 |

#### INTRODUCTION

# Description

This Statistical Analysis Plan (SAP) is consistent with Amendment 4 of the study protocol (dated 2 February 2021) and includes the latest details of efficacy and safety summaries to be included in the clinical study report (CSR).

The preparation of this SAP was done in accordance with STATKING Clinical Services SOP SCI 02-54, Statistical Analysis Plans.

# 1.0 Synopsis of Study Design/Procedures

This study is a prospective, open-label, multicenter, evaluation of the reliability and sensitivity of Tilmanocept Uptake Value (TUV) assessments based on planar imaging localization of intravenously (IV) injected Tc 99m tilmanocept to skeletal joints in subjects with and without active rheumatoid arthritis (RA).

The study has three arms. Arm 1 consists of Healthy Control (HC) subjects. Arm 2 consists of RA patients on stable therapy. Arm 3 consists of RA patients who are candidates for initiation of, or change to a new anti-tumor necrosis factor  $\alpha$  (TNF $\alpha$ ) biological disease-modifying antirheumatic drug (bDMARD) treatment.

The objectives of the study are:

#### **Primary Objectives:**

- To assess the longitudinal precision of TUV<sub>joint</sub> and TUV<sub>global</sub> on planar imaging in subjects with clinically diagnosed active RA on stable antirheumatic therapy.
- To evaluate camera-specific precision of TUV<sub>joint</sub> and TUV<sub>global</sub> on planar imaging in HCs and in subjects with clinically diagnosed active RA using centralized and standardized imaging parameters.
- To assess the correlation of TUV and changes in TUV with changes in clinical assessments at multiple time points after initiation of a new antianti-TNFα bDMARD therapy.

#### Secondary Objectives:

- To assess the temporal post-injection stability of TUV<sub>joint</sub> and TUV<sub>global</sub> at a dose of 150mcg tilmanocept radiolabeled with 10 mCi of Tc 99m.
- To establish normal ranges for TUV<sub>joint</sub> in HCs.

 To assess Tc 99m tilmanocept anatomic localization based on single photon emission computed tomography/ computed tomography (SPECT/CT) imaging of the synovial space in hands and wrists.

# Safety Objective:

 To evaluate safety through the examination of adverse event (AE) incidence and changes over time in laboratory tests, vital signs, and physical examination findings.

## 1.1 Design and Treatment

Subjects will receive the administration of Tc 99m tilmanocept through an IV route of administration. All subjects will receive a 150  $\mu g$  mass dose of tilmanocept labeled with 10 mCi of Tc 99m in a 3 ml volume. Following injection a 10 ml sterile normal saline flush will be administered. The preferred site of IV placement will be between the elbow and wrist.

Arm 1 HC subjects receive a single administration of 10 mCi of Tc 99m in a 150  $\mu g$  mass dose of tilmanocept. Arm 2 RA subjects receive two (2) IV administrations of 10 mCi Tc 99m in a 150  $\mu g$  mass dose of tilmanocept. Arm 3 RA subjects receive up to four (4) administrations of 10 mCi Tc 99m in a 150  $\mu g$  mass dose of tilmanocept.

| Table 1 | Stud | arms |
|---------|------|------|
|---------|------|------|

| Table 1 Study arms | | |
|---|---|---|
| Arm | Subjects | Evaluations |
| 1 | HC subjects clinically free of any inflammatory disease and/or joint pain. | Image, Re-image |
| 2 | Subjects with clinically diagnosed RA who have been on stable anti-rheumatic | Image, Re-image |
| | therapy. | Test, Re-test |
| 3 | Subjects with clinically diagnosed RA who are candidates for initiation of, or change to, a new anti-TNF $\alpha$ bDMARD treatment. | Positive Predictive<br>Value, Negative<br>Predictive Value, |
| | | Clinical Concordance |

#### 1.2 Study Procedures

Subjects will visit the study site for screening procedures up to 30 days (Day -30 to Day -1) before enrollment into the study. Screening procedures (demographics, vital signs, medical history, blood and urine samples for clinical

labs, RA specific labs, urine pregnancy testing for subjects of childbearing potential, and physical exam) will be completed along with RA evaluations using the 2010 ACR/EULAR score. The DAS28 score instrument will be used in Arms 2 and 3.

Subjects arriving for Study Day 0 will be considered enrolled in the study. On Day 0 subjects will receive Tc 99m injection and imaging procedures. Pre-injection procedures include the following: a urine pregnancy test will be administered to all subjects with childbearing potential. Up to 30 minutes prior to drug administration an ECG will be performed, followed by assessment of vital signs and AEs. After pre-injection procedures are completed subjects will receive a single IV dose with 150  $\mu g$  of tilmanocept radiolabeled with 10 mCi of Tc 99m. Within 30 minutes of injection, subjects will receive an ECG followed by vital sign and AE check. Whole body planar imaging will be conducted on the subject at the time points specified for the arm into which he/she was enrolled (see Section 1.0). For subjects in Arms 1 and 2, planar images of the whole body and bilateral hands and wrists will be taken at 60 (± 15) minutes and at 180 (± 15) minutes after injection. Blood will be drawn for clinical laboratory evaluations after all image acquisitions have been completed.

On Study Day 5 ( $\pm$  3 days) a safety follow-up telephone call will include a review of concomitant medications and assessment of adverse events. Arm 1 HC subjects have completed the study at this point.

On Study Day 8 ( $\pm$  1 day) RA subjects in Arm 2 will receive repeat Tc 99m tilmanocept imaging. Pre-injection procedures include the following: a urine pregnancy test will be administered to all subjects with childbearing potential. Up to 30 minutes prior to drug administration an ECG will be performed, followed by assessment of vital signs and AEs. After pre-injection procedures are completed subjects will receive a single IV dose with 150  $\mu$ g of tilmanocept radiolabeled with 10 mCi of Tc 99m. Within 30 minutes of injection, subjects will receive an ECG followed by vital signs and AE assessment. Planar images of the whole body and bilateral hands and wrists will be taken at 60 ( $\pm$  15) minutes and 180 ( $\pm$  15) minutes after injection. Following the 180 minute planar imaging, subjects will have SPECT/CT images of the bilateral hands and wrists taken. Blood will be drawn for clinical laboratory evaluations after all image acquisitions have been completed.

From 1 to 3 days of the second imaging day (i.e., Study Day 9 to 11 if imaging is done on Study Day 8), a safety follow-up telephone call will be made to review concomitant medications and AE check. Arm 2 RA subjects have completed the study at this point.

For RA subjects in Arm 3, Study Day 0 is modified to include planar whole body and planar images of the hands and wrists once only at 60 minutes post-injection. All other procedures remain the same on Study Day 0. The new therapy (anti-

TNF $\alpha$  bDMARD) will be initiated following the Day 0 imaging. A safety follow-up telephone call will be conducted on Study Day 5 (± 3 days). Follow-up images of the hands and wrists and whole body will be made at 5 weeks (± 1 week) after initiation of the new anti-TNF $\alpha$  bDMARD therapy using the same procedures as in Arm 2 Day 8, except that no images will be taken at 180 minutes in Arm 3 and the post imaging clinical laboratory assessments will include an RA panel. CDAI, DAS28, HAQ-DI, WPI, and an AE check will also occur at this visit. A safety follow-up telephone call will be conducted 1 to 3 days later. At weeks 12 (± 1 week) and 24 (± 1 week) after initiation of the new anti-TNF $\alpha$  bDMARD therapy, Arm 3 subjects will have a return visit for imaging and assessment of their RA status. These visits will include clinical laboratory assessments and RA-specific labs (post imaging), tilmanocept injection and image acquisition 60 (± 15) minutes following injection, CDAI, DAS28, HAQ-DI, WPI, and AE check at both of these time points. ACR Response Criteria will be assessed at weeks 5, 12 and 24. After the week 24 visit, Arm 3 RA subjects have completed the study.

The centralized core image laboratory contracted by Navidea Biopharmaceuticals completed a quantitative read of the images to determine the amount of radiotracer uptake in the joints (TUV<sub>joint</sub>) and in the brain (TUV<sub>brain</sub>) for Interim Analysis 2. The core image laboratory will also evaluate localization of Tc 99m tilmanocept in the 180 minute planar and SPECT/CT images of Arm 2 RA patients. Navidea internal work instructions and imaging charter will be followed for all other quantitative and qualitative reads for all other imaging data.

#### 1.3 Sample Size

Up to 105 subjects from up to 10 study centers will be enrolled into Arms 1, 2, and 3 as allocated below, and imaged. Arm 1 will have N = 38 evaluable subjects, Arm 2 will have N = 38 evaluable subjects, and Arm 3 will have N = 29 evaluable subjects. A subject is considered evaluable if he/she meets the criteria for the analysis population and has the data necessary for computing the primary endpoint.

The sample size for Arm 1 was determined to assess temporal stability of the 150  $\mu$ g mass dose/10mCi radiolabeling dose. The sample size for Arm 2 was determined to power a hypothesis test at 0.80:

$$H_0: \pi \le 0.80$$
 $vs$ 
 $H_a: \pi > 0.80$ ,

where  $\pi$  represent the fraction of unsigned differences less than 7.5% The sample size for Arm 3 was determined to provide a lower 97.5% confidence limit for the rank correlation of at most 0.15 when  $\rho$  = 0.70, using Fisher's Z-transformation methods.

# 2.0 Data Analysis Considerations

## 2.1 Types of Analyses

Data analyses described in this SAP will consist of analyzing efficacy and safety data.

## 2.2 Analysis Populations

The following analysis populations will be used in the study:

**Safety Population** – The safety population includes all patients that have been enrolled in the study and injected with at least one dose of Tc 99m tilmanocept.

**Intent-to-Diagnose (ITD) Population** – The ITD population includes all patients that have been enrolled in the study, injected with Tc 99m tilmanocept, and received all imaging and evaluations necessary for the primary endpoint(s) appropriate to their respective arm.

**Per Protocol (PP) Population:** The PP population will include all ITD subjects without major protocol violations. All protocol deviations will be classified as major or minor prior to database lock.

All efficacy analyses will be carried out on the ITD and PP populations with the ITD population being the primary analysis set. All analyses of safety data and baseline subject characteristics will be carried out on the safety population. A data listing displaying the patients excluded from each population will be created, as shown in Appendix B.

#### 2.3 Missing Data Conventions

No missing value imputation will be used in this analysis. All analyses will be based on the observed data.

## 2.4 Interim Analyses

After the injection, imaging, and quantitation of a total of 4 subjects in Arms 1 and 2 combined, an interim analysis (Interim Analysis 1) was held for the review of quantitative TUV results and assessment of imaging parameters and logistics. A second interim analysis was held after a total of 30 subjects (and at least 15 RA subjects) in Arms 1 and 2 were injected, imaged, and quantified for the review of inter- and intra-subject TUV variation to contribute to the power analysis of a future Phase 3 study and/or to terminate the study on grounds of data sufficiency.

After 15 subjects in Arm 3 completed Visit 4, an interim analysis (Interim Analysis 3) was performed to estimate the distribution of treatment effects on TUV and to optimize the TUV metric based on the interim data from all three arms.

Interim analysis plans (IAPs) were written and approved for the second interim analysis of Arms 1 and 2 and for the third interim analysis of all three study arms.

#### 2.5 Calculation of TUV

All calculations are done on a reader-specific basis. That is, there is no statistical aggregation of the reader results.

## **Calculating Joint TUV**

For an individual joint, TUV<sub>joint</sub> is defined as the average pixel intensity of the joint divided by the average pixel intensity of the hand, right or left and anterior or posterior, (includes the region from one wrist region of interest (ROI) diameter above the wrist ROI down to the fingertips).

# **Calculating Global TUV**

For each independent blind reader, determine the average TUV<sub>joint</sub> and 95% prediction interval of both the anterior and posterior views of the wrists, MCPs, and PIPs in healthy individuals (NAV3-31 Arm 1). For all following calculations, reader specific average TUV<sub>joint</sub> and 95% prediction intervals will be used.

For each RA subject do the following.

Step 1: Calculate TUV<sub>joint</sub> for each of the 22 DAS 28 joints for which data are collected.

Step 2: Identify all imaged joints with  $TUV_{joint}$  > upper limit of normal for the anatomically similar joint and view. These will be referred to as inflamed joints (IJ). Each joint has an anterior and posterior view: a joint is considered an IJ if either view has a  $TUV_{joint}$  higher than the upper bound from the normative data set.

Step 3: Calculate the macrophage-involved contribution (MI) to Tc 99m tilmanocept localization for each IJ. This is done by expressing the TUV for the IJ as a fractional change from the mean TUV for the anatomically equivalent joint and view. That is, if  $TUV_{joint}$  and  $\overline{H}_{joint}$  represent the joint and view specific TUV and the mean TUV for the anatomically equivalent joint and view from the normative data set respectively, the macrophage contribution to TUV is  $Ml_{joint}$ :

$$MI_{joint} = \frac{TUV_{joint} - \overline{H}_{joint}}{\overline{H}_{joint}}.$$

Step 4:  $TUV_{global}$  is the total of the macrophage-involved contributions for the IJs. (Note that  $MI_k$  is effectively 0 if  $TUV_{joint}$  is less than or equal to the upper limit of normal from the normative data set.) That is,

$$TUV_{global} = \sum_{All\ IIs} MI_{IJ},$$

$$TUV_{global} = \sum_{k=1}^{22} MI_k.$$

The change in TUV<sub>global[5w]</sub>) is the  $\Delta$ % from baseline (TUV<sub>global[b]</sub>):

$$\Delta TUV_{global[5w]} = 100 \cdot \frac{TUV_{global[5w]} - TUV_{global[b]}}{TUV_{global[b]}}.$$

Arms 1 and 2:

Precision endpoints for both arms will be assessed estimating the mean, standard deviation, n, minimum, median, and maximum of the signed differences (change from baseline) of TUV for each evaluated DAS28 joint. The RMSD will be calculated using the following equation:

$$RMSD = \sqrt{\frac{1}{n-1} \sum_{k=1}^{n} (y_k - w_k)^2}$$

where  $y_k$  and  $w_k$  are the measurements at the two timepoints (for example, the two scans at 60 minutes, the two scans at 180 minutes, or the first 60-minute scan and the first 180-minute scan) and k represents the subject number. A 95% confidence interval for the RMSD based on Normal theory will be provided, as will a 95% bootstrap confidence interval based on N = 5000 bootstrap samples. Box-and-whisker plots of TUV will be provided by arm at each timepoint for each joint, pooling small joints (MCPs and PIPs) and all joints bilaterally. Joints will not be pooled by type or bilaterally in IA 3.

 $\Delta TUV$  will be summarized with descriptive statistics as the signed difference. If  $T_1$  represents the observed TUV at the first time point and  $T_2$  the observed TUV at the second time point, then

$$\Delta TUV = T_2 - T_1.$$

#### Arm 1 Only:

The distribution of TUV<sub>joint</sub> in healthy controls will be summarized by time point for global TUV and each evaluated DAS28 joint with the number of joints, mean, standard deviation, 80<sup>th</sup> and 90<sup>th</sup> percentiles, the median, and 95% prediction limits for a future observation of that type at that time point. Joints will not be pooled. Box-and-whisker plots of the data will be presented by joint and time point. A scatter plot matrix for the three readers will be provided on a joint-specific basis showing the relationship between the reader TUV for the A and B scans.

# Arm 2 Only:

The longitudinal precision of TUV<sub>joint</sub> will be analyzed for each evaluated DAS28 joint. The signed differences will be analyzed with descriptive statistics and the RMSD will be calculated as defined for Arms 1 and 2 above. A 95% confidence interval for the RMSD based on Normal theory will be provided, as will a 95% bootstrap confidence interval based on N = 5000 bootstrap samples. Joints will not be pooled by type or bilaterally. A scatter plot matrix for the three readers will be provided on a joint-specific basis showing the relationship between the reader TUV for the A and B scans.

#### Arm 3 Only:

The Kendall rank correlation between  $\Delta TUV_{global[5w]}$  with  $\Delta CDAI_{12w}$  will be computed and a 95% confidence interval for its value will be computed using Fisher's Z-transformation. Similarly, the Kendall rank correlation between  $\Delta TUV_{global[5w]}$  with changes from baseline in each of the ACR Response Criteria components at 12 weeks (tender joint count (TJC), swollen joint count (SJC), patient assessment of global disease activity, rheumatologist assessment of global disease activity, patient assessment of pain, patient assessment of physical function, and acute-phase reactant value) will be computed and a 95% confidence interval for its value will be computed using Fisher's Z-transformation.

### 2.6 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the control and supervision of the same Principal Investigator (PI). There will be no selective pooling of study centers.

#### 2.7 Documentation and Other Considerations

The data analyses described in this SAP will be conducted using SAS<sup>©</sup> Software, version 9.4 or later.

# 3.0 Analysis of Baseline Patient Characteristics

Baseline and demographic characteristics of the safety population will be summarized by subject arm and overall. Continuous variables (age, height, weight, and time from diagnosis of RA) will be summarized via mean, standard deviation, minimum, maximum, and number of non-missing responses. Categorical variables (gender, race, and ethnicity) will be summarized via counts and percentages.

A detailed listing of baseline data for each patient in the safety population will also be provided, as shown in Appendix B.

# 4.0 Analysis of Efficacy

# 4.1 Description of Efficacy Variables

The efficacy variables for this study are as follows:

- Quantitative determination of TUV<sub>joint</sub> and TUV<sub>global</sub> at Day 0, Day 8, Week 5, Week 12, and Week 24 as appropriate to the subject's study arm.
- Qualitative determination of tilmanocept localization in planar images and SPECT/CT images of the bilateral hands and wrists.
- Subject RA status evaluations in Arm 3 as summarized in the CDAI overall score and its subscores.
- Subject RA status evaluation in Arm 3 as summarized by the ACR Response Criteria.
- Change in TUV.

The presence of radiotracer uptake for a joint indicates the presumed presence of activated macrophages. The use of the term "localization" in this SAP is synonymous with the presence of radiotracer uptake.

TUV is defined as:

$$\mathrm{TUV_{joint}} = \frac{\bar{X}_{joint}}{\bar{X}_{\mathrm{RR}}};$$

where

•  $\bar{X}_{\rm joint}$  is the average voxel intensity of a particular joint of a subject at the anterior or posterior views at 1 or 3-hours post-injection;

•  $\bar{X}_{RR}$  is the average voxel intensity of the reference region (RR) of a subject at the anterior or posterior views at 1 or 3-hours post-injection.

# 4.1.1 Primary efficacy variables

The primary efficacy variables for this study are:

- Quantitative measurement of TUV<sub>joint</sub> (all arms) and TUV<sub>global</sub> (Arms 2 and 3 only)
- CDAI scores at baseline, 12 (± 1) weeks and 24 (± 1) weeks (Arm 3 only)
- DAS28 scores at baseline, 12 (± 1) weeks and 24 (± 1) weeks (Arm 3 only)
- ACR Response Criteria at 12 (± 1) weeks and 24 (± 1) weeks (Arm 3 only).

The primary efficacy variables of this study in Arms 1 and 2 are:

- The camera-specific precision of TUV<sub>joint</sub> and TUV<sub>global</sub> in subjects with active RA and healthy controls, which is defined as the Root Mean Square Difference (RMSD) between the consecutive 15-minute planar images.
- The stability of the mean/variance relationship, which is assessed by comparing the Coefficient of Variation (CV) of TUV<sub>joint</sub> and TUV<sub>global</sub> in subjects with active RA and healthy controls.

An added primary variable in Arm 2 only is:

 The longitudinal (8-day) precision of TUV<sub>joint</sub> and TUV<sub>global</sub> in subjects with active RA, which is defined as the RMSD of the TUV between the baseline and 8 day image at the same time point.

The primary endpoints in Arm 3 are:

- The Kendall rank correlation of  $\Delta TUV_{global[5w]}$  with the response to new anti-TNF $\alpha$  bDMARD therapy defined as  $\Delta CDAl_{12w}$  and  $\Delta CDAl_{24w}$  (overall scores only) in study arm 3.
- The Kendall rank correlation of  $\Delta TUV_{global[5w]}$  with the response to new anti-TNF $\alpha$  bDMARD therapy defined as the changes from baseline in DAS28 and in each of the ACR Response Criteria components at 12 ( $\pm$  1) weeks and at 24 ( $\pm$  1) weeks in study arm 3.

## 4.1.2 Secondary efficacy variables

- Qualitative evaluations of SPECT/CT image detecting localization of Tc 99m tilmanocept in the synovial spaces of the bilateral hands and wrists. (Arm 2 only).
- CDAI score at baseline (CDAI<sub>0w</sub>), 12 (CDAI<sub>12w</sub>) and 24 weeks (CDAI<sub>24w</sub>) (Arm 3 only).
- ACR Response Criteria at 12 and 24 weeks (Arm 3 only).
- Constituent scores of the ACR Response Criteria at baseline, 12 weeks, and 24 weeks, including:
  - o TJC
  - o SJC
  - Patient assessment of global disease activity
  - Rheumatologist assessment of global disease activity
  - Patient assessment of pain
  - Patient assessment of physical function
  - Acute-phase reactant value.
- Constituent scores of the CDAI score
  - o TJC
  - o SJC
  - Patient Global Assessment
  - Physician Global Assessment.

The secondary efficacy endpoints for this study are:

#### ARMS 1-2

• The temporal stability of TUV<sub>joint</sub> and TUV<sub>global</sub> using a 150 mcg tilmanocept mass dose/10 mCi radiolabeling dose, which is defined as the squared difference between the 1-hour and 3-hour planar images. (This endpoint was analyzed to the sponsor's satisfaction in IA-3.)

#### ARM 1

- The normal upper limit of TUV<sub>joint</sub> in HC subjects, which is defined the upper limit of a 95% prediction interval at 60 ±15 minutes:
  - TUV<sub>joint</sub> of evaluated joints (i.e., wrists, MCPs, PIPs, knees, elbows, shoulders in Arms 1 and 2, and wrists, MCPs, and PIPs in Arm 3).

#### ARM 2

• The qualitative evaluations of SPECT/CT in detecting localization within synovial spaces of the bilateral hands and wrists.

#### ARM 3

- TUV<sub>global[0w]</sub> and response to new anti-TNFα bDMARD therapy defined by the change from baseline (CFB) of CDAI to 12 ± 1 weeks and 24 ± 1 weeks (ΔCDAI<sub>12w</sub> and ΔCDAI<sub>24w</sub>, respectively) and by the changes from baseline in each of the ACR Response Criteria components at 12 (± 1) weeks and at 24 (+ 1) weeks.
- $\Delta TUV_{global[5w]}$  and response to new anti-TNF $\alpha$  bDMARD therapy defined by the CFB of CDAI to 12 ± 1 weeks and 24 ± 1 weeks ( $\Delta CDAI_{12w}$  and  $\Delta CDAI_{24w}$ , respectively).
- ΔTUV<sub>global[12w]</sub> and ΔTUV<sub>global[24w]</sub>.
- Concordance of improvement classification using ΔTUV<sub>global[5w]</sub> and ΔTUV<sub>global[5w]</sub> with anti-citrullinated protein/peptide antibody (ACPA) bucketing improvement classification using clinical criteria, including ACR Response Criteria, CDAI, DAS28, and HAQ-DI. See section 4.2.2 below for the definitions of improvement on these clinical criteria.
- Concordance of improvement classification using ΔTUV<sub>global[12w]</sub> and ΔTUV<sub>global[12w]</sub> with ACPA bucketing improvement classification using clinical criteria, including ACR Response Criteria, CDAI, DAS28, and HAQ-DI.
- Response to new anti-TNFα bDMARD therapy defined by the CFB of CDAI to 12 ± 1 weeks and 24 ± 1 weeks (ΔCDAI<sub>12w</sub> and ΔCDAI<sub>24w</sub>, respectively).
- The correlation of ΔTUV<sub>global[5w]</sub> and response to new anti-TNFα bDMARD therapy from baseline to 24 ± 1 weeks defined by the changes from baseline in each of the ACR Response Criteria components.
- Constituent parameters of CDAI<sub>12w</sub>, CDAI<sub>24w</sub>, ΔCDAI<sub>12w</sub>, ΔCDAI<sub>24w</sub>, ACR Response Criteria at 12 and 24 weeks, including:
  - o TJC
  - o SJC
  - Patient assessment of global disease activity
  - Rheumatologist assessment of global disease activity
  - o Patient assessment of pain
  - o Patient assessment of physical function
  - Acute-phase reactant value.

# 4.2 Analysis of Efficacy Variables

## 4.2.1 Primary Efficacy Variables

## Primary Endpoints for Arms 1 and 2

All TUV data will be analyzed with summary statistics (mean, standard deviation, n, minimum, median, maximum) by study arm and joint.

Precision endpoints will be assessed estimating the mean, standard deviation, n, minimum, median, and maximum of the signed differences (CFB). The RMSD will be calculated

$$RMSD = \frac{1}{n-1} \sum_{k=1}^{n} (y_k - w_k)^2$$

where  $y_k$  and  $w_k$  are the measurements at the two timepoints and k represents the subject number. A 95% confidence interval for the RMSD based on Normal theory will provided, as will a 95% bootstrap confidence interval based on N = 5000 bootstrap samples. Timepoints analyzed in this way will include the 60 minute A and B scans, the 180 minute A and B scans, and the difference between the 60 and 180 minute A scans. These will be done for all joints assessed and for TUV<sub>global</sub>. (These analyses were completed to the sponsor's satisfaction in IA-3.)

## Primary Endpoint for Arm 2 Only

The longitudinal (8-day) variation of TUV will be analyzed for each DAS28 joint and globally. The signed differences will be analyzed with descriptive statistics and the RMSD will be calculated as defined for Arm 2 above. A 95% confidence interval for the RMSD based on Normal theory will provided, as will a 95% bootstrap confidence interval based on N = 5000 bootstrap samples will be computed, and 95% confidence limits for its value will be provided. This will be done for TUV<sub>joint</sub> for all evaluated joints and TUV<sub>global</sub> in the 60 minute images using the "A" image at baseline. The fraction of unsigned  $\Delta TUV_{global}$  values less than 7.5% will be summarized in a frequency table and an exact binomial test of the hypotheses described in Section 1.3 will be included for each timepoint.

#### Primary Endpoints for Arm 3 Only

The Kendall rank correlation between  $\Delta TUV_{global[5w]}$  with  $\Delta CDAI_{12w}$  and  $\Delta CDAI_{24w}$  will be computed and a 95% confidence interval for its value will be computed using Fisher's Z-transformation. Similarly, the Kendall rank correlation between  $\Delta TUV_{global[5w]}$  with changes from baseline in DAS28 and in each of the ACR Response Criteria components at weeks 12 and 24 will be computed and a 95% confidence interval for its value will be computed using Fisher's Z-transformation. The marginal distributions of the variables will be characterized with the mean, standard deviation, and the number of data pairs.

# 4.2.2 Secondary Efficacy Variables

# Secondary Endpoints for Arm 1 only

The normal ranges of TUV<sub>joint</sub> will be estimated from data collected from healthy subjects (study arm 1) at 60 minutes post-injection. The mean, standard deviation, n (number of joints), and quantile regression estimates of the 5 and 95 percentiles will be provided for shoulder, elbow, wrist, MCP, PIP, and knee. All joints will be summarized individually.

## Secondary Endpoints for Arms 1 and 2

The temporal quantitative stability of the images will be assessed by computing the fraction of observations for which  $|\Delta TUV_{global}| \le 0.075$  for the difference between the 60 and 180 minute images. The hypotheses

$$H_0: \pi \le 0.80$$

$$vs$$

$$H_a: \pi > 0.80,$$

where  $\pi$  represent the fraction of unsigned differences less than 7.5% will be tested with an exact test and a Clopper-Pearson (exact) 95% confidence interval for p will be provided. The RMSD will be analyzed by joint, providing 95% confidence intervals for the RMSD using both Normal theory methods and a bootstrap estimate with 5000 bootstrap replications.

The 80<sup>th</sup> and 90<sup>th</sup> percentiles of the distribution of unsigned differences will be estimated using quantal regression methods. (These analyses were completed to the sponsor's satisfaction in IA-3.)

#### Secondary Endpoint for Arm 2 only

Qualitative evaluations of SPECT/CT imaging in localizing tilmanocept uptake will be estimated from the active RA subjects (Arm 2 only) on the joints of the hands and wrists. A frequency table of counts and percent of subjects will be provided.

#### Secondary Endpoints for Arm 3 only

All RA quantitative assessment variables (CDAI, ACR Response Criteria component scores, DAS28 score, and HAQ-DI) will be summarized by arm, computing the mean, standard deviation, number of observations, minimum, median, and maximum for the observed values at each time point and for the change from baseline for values collected after Day 0. The ACR Response Criteria will be summarized with a frequency table of the highest ACR Response level (None, ACR20, ACR50, ACR70) attained by that subject at that time point. That is, a subject who satisfies ACR50 also satisfies ACR20 but will not appear in the frequency count for ACR20.

The Kendall rank correlation between  $\Delta TUV_{global}$  at 5 weeks,  $\Delta TUV_{global}$  at 12 and 24 weeks with the component parameters of  $\Delta CDAI_{12w}$  and  $\Delta CDAI_{24w}$  will be computed and 95% confidence intervals for the values provided using Fisher's Z-transformation. This analysis will be repeated for the correlation between  $\Delta TUV_{global}$  at 12 and 24 weeks with change in DAS28 and with ACR Response Criteria components at 12 weeks and 24 weeks (Note: the Kendall rank correlation analysis with DAS28 and ACR Response Criteria components at 5 weeks is a primary endpoint, as described above in Section 4.2.1). The marginal distributions of the variables will be characterized with the mean, standard deviation, and the number of data pairs.

Concordance of improvement classification for: 1)  $\Delta TUV_{global[5w]}$  bucketing; 2)  $\Delta TUV_{global[5w]}$ ; 3)  $\Delta TUV_{global[5w]}$  bucketing with ACPA bucketing; 4)  $\Delta TUV_{global[12w]}$  bucketing; 5)  $\Delta TUV_{global[12w]}$ ; 6)  $\Delta TUV_{global[12w]}$  bucketing with ACPA bucketing; and 7) ACPA bucketing alone with clinical criteria (ACR Response, CDAI, DAS28, and HAQ-DI) will be analyzed as follows.

ACR Response is derived through a combination of reductions from baseline in swollen or tender joint counts as well as improvement from baseline in at least at least 3 of the other parameters (patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant [ESR]). This study will evaluate the following three levels of ACR Response:

- ACR20: An ACR20 indicates that 20% improvement is observed in tender or swollen joint counts as well as 20% improvement in at least 3 of the other 5 criteria.
- ACR50: An ACR50 indicates that 50% improvement is observed in tender or swollen joint counts as well as 50% improvement in at least 3 of the other 5 criteria.
- ACR70: An ACR70 indicates that 70% improvement is observed in tender or swollen joint counts as well as 70% improvement in at least 3 of the other 5 criteria.

Each subject will be classified as a yes or a no for whether they meet each of the above ACR Response Criteria at each of the applicable post-baseline time points. Note that the above criteria are nested, such that if a subject is a yes for ACR70 at a given time point, then the subject is also a yes for ACR50 and ACR20 for that same time point.

A subject will be classified as improved on the CDAI depending on the baseline score as follows:

• If the baseline value is greater than 22, a reduction of more than 12 will be classified as improved. Otherwise, the subject is not improved.

- If the baseline value is between 10 and 22 (inclusive) a decrease of more than 6 will classified as improved. Otherwise, the subject is not improved.
- If the baseline value is less than 10, a decrease of more than 1 will be classified as improved. Otherwise the subject is not improved.

A subject will be classified as improved on the DAS28 with a score change of greater than 1.2.

A decrease of at least 0.22 in the HAQ-DI will be classified as improved. Otherwise, the subject is not improved on the HAQ-DI.

The  $\Delta TUV_{global[5w]}$  values will be used to predict improvement at 12 and 24 weeks according to algorithms 1-3. The  $\Delta TUV_{global[12w]}$  values will be used to predict improvement at 24 weeks according to algorithms 4-6. A seventh algorithm based on ACPA bucketing alone with also be applied to predict improvement at 12 and 24 weeks. Algorithms 1-6 will be applied after the change in TUV calculations have been rounded to the nearest integer percentage (i.e., nearest hundredths place for a proportion).

# 1. ΔTUV<sub>global[5w]</sub> bucketing

In the below, TUV<sub>global</sub> represents the global TUV at the current time point and TUV<sub>global[Day 0]</sub> represents the global TUV at baseline:

- If TUV<sub>global[Day 0]</sub> is < 5 then the prediction is N (No improvement)
- Else if

$$\Delta TUV_{global[5w]} = \frac{TUV_{global[5w]} - TUV_{global[Day0]}}{TUV_{global[Day0]}} \leq -0.10$$

the prediction is Y (patient has improved). That is, a patient will be predicted as improved if  $TUV_{global}$  goes down by greater than or equal to 10%.

Otherwise, the prediction is N.

#### 2. ∆TUV<sub>global[5w]</sub>

The TUV<sub>global</sub> prediction of improvement will also be computed according to the following algorithm:

- If TUV<sub>global</sub> goes down by greater than or equal to 10%, then predict response
- If TUV<sub>global</sub> does not go down by 10% or more, then predict no response
- 3. \( \Delta TUV\_{global[5w]} \) bucketing with ACPA bucketing

The TUV<sub>global</sub> prediction of improvement will also be evaluated by combination of the above two algorithms such that:

For patients with TUV<sub>global</sub> of below 5.0 at baseline:

- ACPA Levels before initiation (at baseline) of the new anti-TNF therapy:
  - ACPA levels ≤85 predicts treatment failure (non-response)
  - ACPA level >85 predicts treatment success (significant clinical improvement)

For patients with TUV<sub>global</sub> at or above 5.0 at baseline:

- If TUV<sub>global</sub> goes down by greater than or equal to 10%, then predict response (no need to refer to ACPA)
- If TUV<sub>global</sub> does not go down by 10% or more, then refer to baseline ACPA for prediction:
  - ACPA levels ≤85 predicts treatment failure (non-response)
  - ACPA level >85 predicts treatment success (significant clinical improvement)

#### 4. ΔTUV<sub>global[12w]</sub> bucketing

In the below, TUV<sub>global</sub> represents the global TUV at the current time point and TUV<sub>global[Day 0]</sub> represents the global TUV at baseline:

- If TUV<sub>global[Day 0]</sub> is < 5 then the prediction is N (No improvement)
- Else if

$$\Delta TUV_{global[12w]} = \frac{TUV_{global[12w]} - TUV_{global[Day0]}}{TUV_{global[Day0]}} \le -0.10$$

the prediction is Y (patient has improved). That is, a patient will be predicted as improved if  $TUV_{global}$  goes down by greater than or equal to 10%.

Otherwise, the prediction is N.

#### 5. ∆TUV<sub>global[12w]</sub>

The TUV<sub>global</sub> prediction of improvement will also be computed according to the following algorithm:

- If TUV<sub>global</sub> goes down by greater than or equal to 10%, then predict response
- If TUV<sub>global</sub> does not go down by 10% or more, then predict no response

## 6. ΔTUV<sub>global[12w]</sub> bucketing with ACPA bucketing

The TUV<sub>global</sub> prediction of improvement will also be evaluated by combination of the above two algorithms such that:

For patients with TUV<sub>global</sub> of below 5.0 at baseline:

- ACPA Levels before initiation (at baseline) of the new anti-TNF therapy:
  - ACPA levels ≤85 predicts treatment failure (non-response)
  - ACPA level >85 predicts treatment success (significant clinical improvement)

For patients with TUV<sub>global</sub> at or above 5.0 at baseline:

- If TUV<sub>global</sub> goes down by greater than or equal to 10%, then predict response (no need to refer to ACPA)
- If TUV<sub>global</sub> does not go down by 10% or more, then refer to baseline ACPA for prediction:
  - ACPA levels ≤85 predicts treatment failure (non-response)
  - ACPA level >85 predicts treatment success (significant clinical improvement)

# 7. ACPA bucketing alone

The following will be used to predict improvement solely on the basis of ACPA:

- ACPA baseline level ≤85 predicts treatment failure (non-response)
- ACPA baseline level >85 predicts treatment success (significant clinical improvement)

For each of the RA improvement criteria, a cross-classification table will be provided. The Uncertainty coefficient for the clinical criterion given the  $\Delta TUV_{\text{global[5w]}}$  of  $\Delta TUV_{\text{global[12w]}}$  classification and its standard error will be calculated. The positive predictive value (PPV), negative predictive value (NPV), and overall accuracy (OA) will be calculated and 95% exact (Clopper-Pearson) confidence intervals will be provided.

PPV and NPV will be calculated as follows, where  $\Delta TUV_{global[xxw]}$  is either  $\Delta TUV_{global[5w]}$  or  $\Delta TUV_{global[12w]}$ , as appropriate:

| Clinical | l Criterion | Classific | ration |
|------------|-------------|-----------|--------|
| Cili iiCai | | Classilic | Jauon |

| $\DeltaTUV_{global[XXw]}$ and/or | | | |
|----------------------------------|------------------|--------------|---------|
| ACPA Classification | Improved | Not Improved | Total |
| Improved | Α | В | A+B |
| Not Improved | С | D | C+D |
| Total | A+C | B+D | A+B+C+D |
| | PPV = A/(A) | A+B) | |
| | NPV = D/( | C+D) | |
| | OA = (A+D)/(A-C) | +B+C+D). | |

A separate table will be provided to summarize the baseline ACPA levels on a continuous scale and the number and percentage of subjects in each ACPA category ( $\leq$ 70, >70).

Figures displaying the  $\Delta TUV_{global}$  by time point (5, 12, and 24 weeks) will be created to display the relationship between  $\Delta TUV_{global}$  over time with the corresponding clinical response assessment (ACR20/50/70, DAS28, and CDAI) at the given time point.

# 5.0 Analysis of Safety

# 5.1 Description of Safety Variables

The safety analysis variables are defined as follows:

- Adverse Events (AEs)
- Clinical Laboratory Tests (hematology, serum chemistry, urinalysis, RA panel)
- ECG Parameters
- Vital Signs

#### 5.2 Description of Safety Analysis

The following describes the safety analyses to be performed for the study. All safety analyses will be performed on the safety population. Follow up timing will vary by arm as noted above.

#### **Adverse Events**

Adverse events will be observed for each subject from signing of informed consent until termination from the study. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®). A treatment-emergent AE (TEAE) is defined as an AE whose start date is on or after the initial procedure date. Based on the coded terms, frequencies of each TEAE will be summarized

by MedDRA® preferred term within system organ class (SOC), by severity grade, and by relationship to Tc 99m Tilmanocept for each arm and overall.

A summary of TEAEs will be constructed showing the following by arm and overall:

- Number of subjects with at least one TEAE
- TEAEs by arm and severity grade
- TEAE by arm and relationship to Tc 99m tilmanocept
- TEAEs by arm and relationship of TEAE to study procedure
- Number of subjects with at least one treatment emergent serious adverse event

Treatment-emergent serious adverse events (TESAEs) will be tabulated by MedDRA® preferred term within SOC by arm and overall.

A by-patient AE data listing of all AEs including verbatim term, coded term, grade, and relation to study drug will be provided.

# **Clinical Laboratory Tests**

Clinical laboratory tests will be performed at screening (baseline) and after the final image acquisition on each imaging day. Only abnormal laboratory values and RA lab values will be assessed for clinical significance as applicable. For each quantitative laboratory test, summary statistics (mean, standard deviation, median, range, n) on the raw as well as their changes from baseline will be presented by timepoint by arm and overall. A shift table will also be produced to show the changes in lab values over time relative to the normal ranges.

If multiple labs were performed at a given visit, then the latest results will be summarized in the analysis tables. All collected lab data will be listed.

#### **ECG Parameters**

ECGs will be performed just prior and just after injection. For each ECG parameter (heart rate, QRS, QT, PR, and QTcF), summary statistics (mean, standard deviation, median, range, n) on the raw as well as their changes from baseline will be presented by timepoint, by arm, and overall. A shift table will be provided to show changes in the qualitative assessment (abnormal or normal) from baseline (pre-injection) to post-injection. The baseline value for each of the post-injection ECG parameters will be the corresponding pre-injection time point. All ECG data will be listed.

#### Vital Signs

Vital signs will be performed at screening, just prior to and just after injection. Height and weight will be measured only at screening and will be summarized as part of the baseline and demographic information. For each vital sign (respiration

rate, systolic blood pressure, diastolic blood pressure, heart rate and temperature), summary statistics (mean, standard deviation, minimum, maximum, n) on the raw as well as their changes from baseline will be presented by timepoint, by dose, and overall. The baseline value for each of the post-injection vital sign parameters will be the corresponding pre-injection time point. If there are multiple vital signs taken at any time point, then the latest set of vital signs will be used for the analysis. All vital sign data will be listed.

# 6.0 Other Relevant Data Analyses/Summaries

# **6.1 Patient Completion**

A table will be constructed with counts of screen failures and enrolled subjects. Of those enrolled, counts and percentages of patients withdrawing from the study before study completion and the number completing the study will be displayed. For those subjects that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. The table will include summary counts and percentages by study arm and overall. A data listing of all subject completion and withdrawal data will also be constructed.

# 6.2 Physical Exam

Physical exams will be performed at screening. All physical exam data will be listed.

# 6.3 Study Drug Administration

The volume, the calculated mass dose, and radioactivity of Tc 99m Tilmanocept injected will be summarized by arm and overall. All study drug administration data will be listed.

# 6.4 RA Evaluation and Screening Physical Exam

Each RA subject will undergo a DAS28 evaluation during screening. Arm 3 subjects will also undergo a DAS28 evaluation at weeks 5, 12, and 24. The swollen and tender joints will be identified and documented during the physical examination. Results of all DAS28 evaluations will be listed.

#### 6.5 Concomitant Medications

All prior and concomitant medications will be listed, as shown in Appendix B. A separate data listing will be created to show only those medications that were taken for RA within the 6 months prior to Day 0 injection. In addition to the summarization of prior RA-specific treatments, recent or concomitant treatments

taken for RA in the last 6 months must be collected in accordance with the following time windows:

- Traditional DMARDs: On therapy at least 90 days and at a stable dose at least 30 days prior to the first imaging visit (Day 0)
- bDMARDs: More than 180 days prior to the first imaging visit (Day 0)
- JAK inhibitors: More than 180 days prior to the first imaging visit (Day 0)
- NSAIDs/Corticosteroids: At least 28 days prior to the first imaging visit (Day 0)

# 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included in Final Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 1 | Subject Disposition by Study Arm | X | X |
| 2 | Demographics and Baseline Data Summary Statistics by Arm - Continuous Variables (Safety Population) | Х | Х |
| 3 | Demographics and Baseline Data Summary Statistics by Arm – Categorical Variables (Safety Population) | X | X |
| 4 | Summary of Study Drug Administration by Arm (Safety Population) | Х | Х |
| 5 | Summary of TUV by Arm, Study Day, and DAS28 Joint (ITD population) | Х | Х |
| 6 | Summary of TUV by Arm, Study Day, and DAS28 Joint (PP Population) | Х | |
| 7 | Summary for Eight-Day Longitudinal Stability of TUV (Arm 2 Only) (ITD Population) | Х | Х |
| 8 | Summary for Eight-Day Longitudinal Stability of TUV (Arm 2 Only) (PP Population) | Х | |
| 9 | Analysis of Eight-Day Longitudinal Stability of ∆TUV <sub>global</sub> (ITD population) | Х | Х |
| 10 | Analysis of Eight-Day Longitudinal Stability of ∆TUV <sub>global</sub> (PP population) | Х | Х |
| 11 | Summary for Day 0 vs Day 8 RA Images (ITD Population) | Х | Х |
| 12 | Summary for Day 0 vs Day 8 RA Images (PP Population) | X | |
| 13 | Assessment of Mean/Variance Relationship by Time Point (ITD Population) | X | X |
| 14 | Assessment of Mean/Variance Relationship by Time Point (PP Population) | Х | |
| 15 | Normal Range of TUV in Healthy Control Subjects (ITD Population) | Х | Х |
| 16 | Normal Range of TUV in Healthy Control Subjects (PP Population) | Х | |
| 17 | RA Status Summaries (ITD Population) | Х | Х |
| 18 | RA Status Summaries (PP Population) | X | |
| 19 | Kendall Rank Correlation of $\Delta TUV$ , $\Delta CDAI$ , $\Delta ACR$ Response Criteria Components, and $\Delta DAS28$ with $\Delta TUV$ at 5 weeks in Arm 3 (ITD Population) | Х | X |
| 20 | Kendall Rank Correlation of ΔTUV, ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 5 weeks in Arm 3 (PP Population) | Х | |
| 21 | Kendall Rank Correlation of ΔTUV, ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 12 weeks in Arm 3 (ITD Population) | Х | Х |
| 22 | Kendall Rank Correlation of ΔTUV, ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 12 weeks in Arm 3 (PP Population) | Х | |

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 23 | Kendall Rank Correlation of ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 24 weeks in Arm 3 | X | X |
| 24 | (ITD Population) Kendall Rank Correlation of ΔCDAI, ΔACR Response Criteria Components, and ΔDAS28 with ΔTUV at 24 weeks in Arm 3 (PP Population) | Х | |
| 25 | Frequency Counts of Localization in SPECT/CT Imaging in RA-2 Subjects (ITD Population) | Х | Х |
| 26 | Frequency Counts of Localization in SPECT/CT Imaging in RA-2 Subjects (PP Population) | Х | |
| 27 | Number and Percentage of Subjects with TEAEs (Safety Population) | Х | Х |
| 28 | Summary of TEAEs (Safety Population) | Х | Х |
| 29 | Number and Percentage of Subjects with TESAEs (Safety Population) | X | X |
| 30 | Number and Percentage of Subjects With TEAEs by Severity Grade (Safety Population) | Х | Х |
| 31 | Number and Percentage of Subjects With TEAEs by Level of Relationship to Tc 99m Tilmanocept (Safety Population) | Х | |
| 32 | Number and Percentage of Subjects With TEAEs by Level of Relationship to Procedure (Safety Population) | Х | Х |
| 33 | Serum Chemistry Clinical Laboratory Parameters Summary<br>Statistics by Arm (Safety Population) | Х | Х |
| 34 | Hematology Clinical Laboratory Parameters Summary<br>Statistics by Arm (Safety Population) | Х | |
| 35 | Urinalysis Clinical Laboratory Parameters Summary Statistics by Arm (Safety Population) | Х | |
| 36 | Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm (Safety Population) | Х | Х |
| 37 | Hematology Clinical Laboratory Parameters Shift Table by Arm (Safety Population) | Х | |
| 38 | Urinalysis Clinical Laboratory Parameters Shift Table by Arm (Safety Population) | Х | |
| 39 | ECG Parameters Summary Statistics by Arm (Safety Population) | Х | Х |
| 40 | ECG Shift Table by Arm (Safety Population) | Х | Х |
| 41 | Vital Signs Summary Statistics by Arm (Safety Population) | Х | Х |
| 42 | ACR Response Classification by Time Point (ITD Population) | Х | Х |
| 43 | ACR Response Classification by Time Point (PP Population) | Х | |
| 44 | Concordance of $\Delta TUV_{global[5w]}$ Bucketing and Week 12 Clinical Improvement Criteria (ITD Population) | X | X |
| 45 | Concordance of ΔTUV <sub>global[5w]</sub> Bucketing and Week 12 Clinical Improvement Criteria (PP Population) | Х | |
| 46 | Concordance of ΔTUV <sub>global[5w]</sub> Bucketing and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 47 | Concordance of $\Delta TUV_{global[5w]}$ Bucketing and Week 24 Clinical Improvement Criteria (PP Population) | X | |
| 48 | Concordance of ΔTUV <sub>global[5w]</sub> and Week 12 Clinical Improvement Criteria (ITD Population) | Х | |

| Table<br>No. | Table Title | Included in Final Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 49 | Concordance of ∆TUV <sub>global[5w]</sub> and Week 12 Clinical Improvement Criteria (PP Population) | X | |
| 50 | Concordance of ∆TUV <sub>global[5w]</sub> and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 51 | Concordance of ΔTUV <sub>global[5w]</sub> and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 52 | Concordance of $\Delta TUV_{global[5w]}$ Bucketing with ACPA Bucketing and Week 12 Clinical Improvement Criteria (ITD Population) | Х | |
| 53 | Concordance of $\Delta TUV_{global[5w]}$ Bucketing with ACPA Bucketing and Week 12 Clinical Improvement Criteria (PP Population) | Х | |
| 54 | Concordance of $\Delta TUV_{global[5w]}$ Bucketing with ACPA Bucketing and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 55 | Concordance of $\Delta TUV_{global[5w]}$ Bucketing with ACPA Bucketing and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 56 | Concordance of ΔTUV <sub>global[12w]</sub> Bucketing and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 57 | Concordance of ΔTUV <sub>global[12w]</sub> Bucketing and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 58 | Concordance of ΔTUV <sub>global[12w]</sub> and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 59 | Concordance of ΔTUV <sub>global[12w]</sub> and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 60 | Concordance of ΔTUV <sub>global[12w]</sub> Bucketing with ACPA Bucketing and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 61 | Concordance of $\Delta TUV_{global[12w]}$ Bucketing with ACPA Bucketing and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 62 | Concordance of ACPA Bucketing Alone and Week 12 Clinical Improvement Criteria (ITD Population) | Х | |
| 63 | Concordance of ACPA Bucketing Alone and Week 12 Clinical Improvement Criteria (PP Population) | Х | |
| 64 | Concordance of ACPA Bucketing Alone and Week 24 Clinical Improvement Criteria (ITD Population) | Х | |
| 65 | Concordance of ACPA Bucketing Alone and Week 24 Clinical Improvement Criteria (PP Population) | Х | |
| 66 | ACPA Summary Statistics in Arm 3 (ITD Population) | X<br>X | Х |
| 67 | ACPA Summary Statistics in Arm 3 (PP Population) | Х | |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Figures | Shown in<br>Appendix<br>B |
|---|---|---|---|
| Fig1 | Plot of ΔTUV <sub>global</sub> by Imaging Time Point and ACR-20 for Arm 3 (ITD Population) | Х | X |
| Fig2 | Plot of ΔTUV <sub>global</sub> by Imaging Time Point and ACR-50 for Arm 3 (ITD Population) | Х | |
| Fig3 | Plot of ΔTUV <sub>global</sub> by Imaging Time Point and ACR-70 for Arm 3 (ITD Population) | Х | |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Figures | Shown in<br>Appendix<br>B |
|---|---|---|---|
| Fig4 | Plot of $\Delta TUV_{global}$ by Imaging Time Point and CDAI for Arm 3 (ITD Population) | X | |
| Fig5 | Plot of $\Delta TUV_{global}$ by Imaging Time Point and DAS28 for Arm 3 (ITD Population) | Х | |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix<br>B |
|---|---|---|---|
| DL1 | Subject Disposition Data Listing | X | X |
| DL2 | Inclusion/Exclusion Data Listing | X | X |
| DL3 | Protocol Deviations Data Listing | X | X |
| DL4 | Demographics Data Listing | X | X |
| DL5 | Subjects Excluded from ITD Population Data Listing | X | X |
| DL6 | Subjects Excluded from PP Population Data Listing | X | X |
| DL7 | Subjects Excluded from Safety Population Data Listing | X | X |
| DL8 | Medical History Data Listing | X | X |
| DL9 | Prior and Concomitant Medications Data Listing | X | X |
| DL10 | Prior and Concomitant RA Medications Data Listing | X | X |
| DL11 | Adverse Events Data Listing | X | X |
| DL12 | Subject Laboratory Profiles – Hematology Data Listing | X | X |
| DL13 | Subject Laboratory Profiles – Serum Chemistry Data Listing | Х | |
| DL14 | Subject Laboratory Profiles – Urinalysis Data Listing | Х | |
| DL15 | Subject Laboratory Profiles – Rheumatology Panel Data<br>Listing | X | |
| DL16 | Physical Exam Data Listing | Х | X |
| DL17 | ACR/EULAR 2010 Classification Data Listing | Х | X |
| DL18 | ACR Data Listing | Х | X |
| DL19 | CDAI, DAS28, HAQ-DI, and WPI Scores Data Listing | Х | X |
| DL20 | DAS-28 by Joint Data Listing | Х | Х |
| DL21 | DAS-28 by Subject Data Listing | Х | X |
| DL22 | Vital Signs Data Listing | Х | X |
| DL23 | ECG Parameters Data Listing | Х | X |
| DL24 | Study Drug Administration Data Listing | Χ | Х |
| DL25 | Post-Injection Imaging Data Listing | X | X |
| DL26 | SPECT/CT Reader Results Data Listing – Hands and Wrists | X | Х |
| DL27 | TUV Data Listing | X | Х |
| DL28 | ACR Response Criteria Data Listing | Х | Х |

# 9.0 References

Food & Drug Administration Center for Drug Evaluation and Research and Center for Biologics Evaluation and Research (September 1998). Guidance for Industry: ICH E9 Statistical Principles for Clinical Trials.

Forkman, J. (2009) Estimator and Tests for Common Coefficients of Variation in Normal Distributions. *Communications in Statistics: Theory and Methods*. **38**:2, pp233-251.

# **Appendix A – Tables, Figures and Listing Specifications**

#### Orientation

Tables and figures will be displayed in landscape.

## Margins

Margins will be 1 inch on all sides. Table and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### Headers

The table number will be on the first line of the title. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, 1 line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (DD-MMM-YYYY)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

#### **Table Disclaimer**

The format of the mock tables shown in the appendix of this SAP will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.
#### **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

#### **Display of Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (ie, for a missing day value, the value displayed is in yyyy-mm format).

Appendix B – Table Shells

Page x of y

Table 1. Subject Disposition by Study Arm Navidea Biopharmaceuticals - Study No. NAV3-31

| | | Arma | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | HC | | RA-2 | | RA-3 | 70 | verall |
| | | (N | = xx | (N | $=$ $\times \times$ ) | (N | = xx | (N | = xx) |
| Screen Failures | | | | | | | | | XX |
| Enrolled | | | XX | | XX | | XX | | XX |
| Completed | | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| Withdrawn | | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | xx | (xxx%) |
| Withdrawal Reason | Adverse Event<br>Protocol Violation | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Lost to Follow Up | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Withdrawal of Consent | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Sponsor Discretion | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Investigator Discretion | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Death | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Other | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |

<sup>&</sup>lt;sup>a</sup> HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

The denominator for all percentages in the table is the number of enrolled subjects in the respective arm and overall. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 2. Demographics and Baseline Data Summary Statistics by Arm - Continuous Variables

Navidea Biopharmaceuticals - Study No. NAV3-31

Safety Population (N=xxx)

| Variable | Arma | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|
| Age (years) | HC | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | xxx | XXX | XXX | xxx | XXX | XXX |
| | RA-3 | XXX | XXX | XXX | XXX | XXX | XXX |
| Height (inches) | HC | xxx | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | xxx | XXX | XXX | XXX | XXX | XXX |
| Weight (pounds) | HC | xxx | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | xxx | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | xxx | XXX | XXX | XXX | XXX | XXX |
| Time from Diagnosis of RA (months) <sup>b</sup> | RA-2 | XXX | xxx | XXX | XXX | xxx | XXX |
| | RA-3 | XXX | xxx | XXX | XXX | xxx | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

 $<sup>^{</sup>a}$  HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

b Calculated as the difference between date of enrollment and date of RA diagnosis.

Page x of y

Table 3. Demographics and Baseline Data Summary Statistics by Arm - Categorical Variables Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| | | | Arma | |
|---|---|---|---|---|
| | | HC | RA-2 | RA-3 |
| Variable | Category | (N=xxx) | (N=xxx) | (N=xxx) |
| Gender | Male | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Female | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Race | American Indian or Alaska Native | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Asian | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Black or African American | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Native Hawaiian or Other Pacific Islander | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | White | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Other | | | |
| Ethnicity | Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Not Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

 $<sup>^{</sup>a}$  HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 4. Summary of Study Drug Administration by Arm Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| | Arma | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|
| | | | | | | | _ |
| Tc 99m Dose (mCi) | HC | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | RA-2 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | RA-3 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| Mass Dose (μg) | HC | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | RA-2 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | RA-3 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| Total Volume of Tc 99m Tilmanocept Injected (mL) | HC | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | RA-2 | XXXX | xxxx | XX | xxxx | xxxx | XXXX |
| | RA-3 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 5. Summary of TUV by Arm, Study Day and DAS28 Joint
Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Number

| | | | | of | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ${\tt Arm^a}$ | DAS28 Joint | Study Day | View | Subjects | Mean | Std Dev | n | Min | Max | Median |
| | | | | | | | | | | · |
| XXXX | XXXXXXXXXXXXX | XXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | XXXXXXXXXXXXXX | XXXX | XXXXXXXX | XX | xxxx.x | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | XXXXXXXXXXXXXX | XXXX | XXXXXXXX | XX | xxxx.x | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

All evaluated DAS28 joints for all groups (HC, RA-2, RA-3), all imaging days (for RA-2 and RA-3 only). Table format is repeated for the PP population.

 $<sup>^{</sup>a}$  HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

Page x of y

Table 7. Summary for Eight-Day Longitudinal Stability of TUV (Arm 2 Only)

Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 1 of 4

| | | | Number | | | Coefficient | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Global TUV or | | | of | Mean | | of | | | | |
| DAS28 Joint TUV | View | Reader | Subjects | Difference | Std Dev | Variation | n | Min | Max | Median |
| xxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | xx.xx |
| XXXXXXXXXXXXXXX | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XX |
| xxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XX |
| XXXXXXXXXXXXXXX | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XX |
| XXXXXXXXXXXXXXX | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XX |
| XXXXXXXXXXXXXXX | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XX |
| xxxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XX |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 7. Summary for Eight-Day Longitudinal Stability of TUV (Arm 2 Only)

Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 2 of 4

| Global TUV or<br>DAS28 Joint TUV | View | Daadaa | Number<br>of | Mean<br>Absolute | 80 <sup>th</sup> Percentile<br>of Absolute<br>Differences | 90 <sup>th</sup> Percentile<br>of Absolute |
|---|---|---|---|---|---|---|
| DAS28 JOINT TOV | view | Reader | Subjects | Difference | Differences | Differences |
| XXXXXXXXXXXXXX | XX | XX | XX | XX.XXX | XX.XX | XX.XX |
| xxxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XX | XX.XX |
| xxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XX | XX.XX |
| XXXXXXXXXXXXXX | XX | XX | XX | xx.xxx | XX.XX | XX.XX |
| xxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XX | XX.XX |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 7. Summary for Eight-Day Longitudinal Stability of TUV (Arm 2 Only)

Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 3 of 4

| | | | Percent | |
|---|---|---|---|---|
| Global TUV or | | | $ \Delta \text{TUV} $ < | 95% Exact |
| DAS28 Joint TUV | View | Reader | 7.5% | Confidence Limits |
| xxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) |
| xxxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) |
| xxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) |
| xxxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) |
| xxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) |
| xxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) |
| xxxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 7. Summary for Eight-Day Longitudinal Stability of TUV (Arm 2 Only)

Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 4 of 4

| Global TUV or | | | | 95% Confidence | 95% Bootstrap |
|---|---|---|---|---|---|
| DAS28 Joint TUV | View | Reader | RMSD | Limits | Confidence Limits |
| xxxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 9. Analysis of Eight-Day Longitudinal Stability of  $\Delta TUV_{global}$  Navidea Biopharmaceuticals - Study No. NAV3-31 ITD Population (N=xxx)

| | | | | 95% Exact | |
|---|---|---|---|---|---|
| Reader | $ \Delta TUV_{global} \leq 7.5\%$ | Frequency | Fraction | Confidence Limits | P-value <sup>1</sup> |
| XXX | True | xx | x.xxx | (x.xxx, x.xxx) | x.xxxx |
| *** | False | XX | x.xxx | (x.xxx, x.xxx) | A.XXXX |
| | 14150 | AA | A.AAA | | |
| XXX | True | XX | X.XXX | (x.xxx, x.xxx) | x.xxxx |
| | False | XX | x.xxx | | |
| XXX | True | XX | X.XXX | (x.xxx, x.xxx) | X.XXXX |
| | False | XX | X.XXX | | |

Source Program: xxxxxxx.sas

Table format is repeated for the PP population.

 $<sup>^1</sup>$  Exact binomial test of the hypotheses  $H_0\colon\,\pi\,\leq\,0.80$  vs  $H_1\colon\,\pi\,>\,0.80$  . STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 11. Summary of Day 0 vs Day 8 RA Images
Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 1 of 2

Standard Deviation

| | | | | | Deviacion | | | |
|---|---|---|---|---|---|---|---|---|
| Global TUV or | | | Number of | Mean | of | Minimum | Median | Maximum |
| DAS28 Joint TUV | View | Reader | Joints | Difference | Difference | Difference | Difference | Difference |
| xxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XX |
| xxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XX |
| xxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XX |
| xxxxxxxxxxxxx | XX | XX | XX | XX.XXX | XX.XXX | XX.XX | XX.XX | XX.XX |

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 11. Summary of Day 0 vs Day 8 RA Images
Navidea Biopharmaceuticals - Study No. NAV3-31
ITD Population (N=xxx)

Part 2 of 2

| | | | $ \Delta exttt{TUV}_{	exttt{global}} $ | 95% Confidence | | |
|---|---|---|---|---|---|---|
| DAS28 Joint | Reader | View | <u>&lt;</u> 7.5% | Limits | 80 %tile | 90 %tile |
| XXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| xxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| xxxxxxxxxxxx | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |
| XXXXXXXXXXXXXXX | XX | XX | XX.XXX | (xx.xxx, xx.xxx) | XX.XXX | XX.XXX |

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 13. Assessment of Mean/Variance Relationship by Time Point
Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 1 of 2

Number Global TUV or of DAS28 Joint TUV Median View Reader Arma Joints Mean Std Dev Minimum Maximum XXXXXXXXXXXXXX XX XX HC XX XX.XXX XX.XXX XX.XX XX.XX XX.XX RA-2 XX XX.XXX XX.XXX XX.XX XX.XX XX.XX XX HC XXXX.XXX XX.XXX XX.XX XX.XX XX.XX RA-2 XXXX.XXX XX.XXX XX.XX XX.XX XX.XX HC XXXX.XXX XX.XXX XX.XX XX.XX XX.XX RA-2 XX XX.XXX XX.XXX XX.XX XX.XX XX.XX XX HC XX XX.XXX XX.XXX XX.XX XX.XX XX.XX RA-2 xx.xxx xx.xxx XX xx.xx xx.xx xx.xx HС XX XX.XXX XX.XXX XX.XX XX.XX XX.XX XX RA-2 XXXX.XXX XX.XXX XX.XX XX.XX XX.XX HC XX XXXX.XXX XX.XXX XX.XX XX.XX XX.XX RA-2 XX.XXX XX.XXX XX.XX XX.XX XX.XX

BC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen).

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxxx.sas

Page x of y

Table 13. Assessment of Mean/Variance Relationship by Time Point
Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 2 of 2

| | | | | Coefficient | | Bootstrap |
|---|---|---|---|---|---|---|
| Global TUV or | | | | of | 95% Confidence | Confidence |
| DAS28 Joint TUV | View | Reader | ${\tt Arm^a}$ | Variation | Limits | Interval |
| xxxxxxxxxxxx | XX | XX | HC | XX.XXX | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |
| | | | RA-2 | XX.XXX | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |
| | | XX | HC | XX.XXX | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |
| | | | RA-2 | XX.XXX | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |
| | | XX | HC | XX.XXX | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |
| | | | RA-2 | XX.XXX | (xx.xxx, xx.xxx) | (xx.xxx, xx.xxx) |

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen).

Page x of y

Table 15. Normal Range of TUV in Healthy Control Subjects
Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

| | | | Number of | | Standard | Estimated | Estimated |
|---|---|---|---|---|---|---|---|
| Joint | View | Reader | Joints | Mean | Deviation | 5 %tile | 95 %tile |
| xxxxxxxxxx | xx | xx | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |
| | | xx | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |
| | | xx | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |
| | xx | xx | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |
| | | xx | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |
| | | XX | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

DAS28 joints will not be pooled in this table. Table format is repeated for the PP population.

Page x of y

# Table 17. RA Status Summaries Navidea Biopharmaceuticals - Study No. NAV3-31 ITD Population (N=xxx)

| Arma | RA Status<br>Measure | Study<br>Visit | Data<br>Type | Mean | Standard<br>Deviation | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxxxxxxxx | xxx | Baseline | xxxx.x | xxx.xx | xxx | xxxx.x | XXXX.X | xxxx.x |
| 21212121 | | XXX | RAW | xxxx.x | xxx.xx | xxx | xxxx.x | xxxx.x | xxxx.x |
| | | | CFB | XXXX.X | xxx.xx | XXX | XXXX.X | XXXX.X | xxxx.x |
| | xxxxxxxxxx | xxx | Baseline | xxxx.x | xxx.xx | xxx | xxxx.x | xxxx.x | xxxx.x |
| | ********** | XXX | RAW | XXXX.X | xxx.xx | XXX | XXXX.X | xxxx.x | XXXX.X |
| | | | CFB | xxxx.x | xxx.xx | xxx | xxxx.x | xxxx.x | xxxx.x |
| | | | Danalina | | | | | | |
| | XXXXXXXXXX | XXX | Baseline<br>RAW | XXXX.X | XXX.XX<br>XXX.XX | XXX | xxxx.x<br>xxxx.x | XXXX.X<br>XXXX.X | xxxx.x<br>xxxx.x |
| | | | CFB | xxxx.x | xxx.xx | xxx | xxxx.x | xxxx.x | xxxx.x |

Table format is repeated for the PP population. RAW and CFB lines will exist only for ARM RA-3.

<sup>&</sup>lt;sup>a</sup> RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 19. Kendall Rank Correlation of  $\Delta$ TUV,  $\Delta$ CDAI,  $\Delta$ ACR Response Criteria Components, and  $\Delta$ DAS28 with  $\Delta$ TUV at 5 Weeks in Arm 3 Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 1 of 3: Reader x

| Measureª | Component<br>Parameter | Time Point | Kendall<br>Correlation <sup>b</sup> | 95% Confidence<br>Limits <sup>c</sup> | n | Mean | Standard<br>Deviation |
|---|---|---|---|---|---|---|---|
| $\Delta$ TUV | | 5 Weeks | | | xxx | xxxxx | xxxxxx |
| $\Delta$ TUV | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | XXXXXX | xxxxxx |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | XXX | XXXXXX | XXXXXX |
| ΔCDAI | Overall | 5 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | XXXXXX |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| ΔCDAI | xxxxxxx | 5 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| ΔACR | xxxxxxx | 5 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | XXXXXX | XXXXXX |
| | | 24 Weeks | X.XXX | (x.xxx, x.xxx) | XXX | XXXXXX | XXXXXX |
| ΔDAS28 | | 5 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |
| | | 12 Weeks | x.xxx | (x.xxx, x.xxx) | XXX | xxxxxx | xxxxxx |
| | | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |

<sup>&</sup>lt;sup>a</sup> Change in ACR will be evaluated through the following components of the ACR Response Criteria: swollen joint count, tender joint count, patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant (ESR).

Source Program: xxxxxxx.sas

Table format is repeated for each reader. Entire table (all parts) is repeated for the PP population.

 $<sup>^{</sup>m b}$  Kendall rank correlation between  $\Delta$ TUV at 5 weeks and the indicated measurement and time point.

<sup>°</sup> Confidence limits calculated using Fisher's Z-transformation.

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 21. Kendall Rank Correlation of  $\Delta$ TUV,  $\Delta$ CDAI,  $\Delta$ ACR Response Criteria Components, and  $\Delta$ DAS28 with  $\Delta$ TUV at 12 Weeks in Arm 3

Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 1 of 3: Reader x

| Measure <sup>a</sup> | Component<br>Parameter | Time Point | Kendall<br>Correlation <sup>b</sup> | 95% Confidence<br>Limits° | n | Mean | Standard<br>Deviation |
|---|---|---|---|---|---|---|---|
| $\Delta$ TUV | | 12 Weeks | | | xxx | xxxxx | xxxxxx |
| ΔΤUV | | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxx | xxxxxx |
| ΔCDAI | Overall | 12 Weeks<br>24 Weeks | x.xxx<br>x.xxx | (x.xxx, x.xxx)<br>(x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| ΔCDAI | xxxxxxx | 12 Weeks<br>24 Weeks | x.xxx<br>x.xxx | (x.xxx, x.xxx)<br>(x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| $\Delta$ acr | xxxxxxx | 12 Weeks<br>24 Weeks | x.xxx<br>x.xxx | (x.xxx, x.xxx)<br>(x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| ∆DAS28 | | 12 Weeks<br>24 Weeks | x.xxx<br>x.xxx | (x.xxx, x.xxx)<br>(x.xxx, x.xxx) | xxx<br>xxx | xxxxxx | xxxxxx |

Source Program: xxxxxxx.sas

Table format is repeated for each reader. Entire table (all parts) is repeated for the PP population.

<sup>&</sup>lt;sup>a</sup> Change in ACR will be evaluated through the following components of the ACR Response Criteria: swollen joint count, tender joint count, patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant (ESR).

 $<sup>^{</sup>m b}$  Kendall rank correlation between  $\Delta$ TUV at 12 weeks and the indicated measurement and time point.

<sup>&</sup>lt;sup>c</sup> Confidence limits calculated using Fisher's Z-transformation.

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 23. Kendall Rank Correlation of  $\Delta$ CDAI,  $\Delta$ ACR Response Criteria Components, and  $\Delta$ DAS28 with  $\Delta$ TUV at 24 Weeks in Arm 3

Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

Part 1 of 3: Reader x

| Measure <sup>a</sup> | Component<br>Parameter | Time Point | Kendall<br>Correlation <sup>b</sup> | 95% Confidence<br>Limits <sup>c</sup> | n | Mean | Standard<br>Deviation |
|---|---|---|---|---|---|---|---|
| ΔΤUV | | 24 Weeks | | | xxx | xxxxxx | xxxxxx |
| ΔCDAI | Overall | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| ΔCDAI | xxxxxxx | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| ΔACR | xxxxxxx | 24 Weeks | x.xxx | (x.xxx, x.xxx) | xxx | xxxxxx | xxxxxx |
| ∆DAS28 | | 24 Weeks | x.xx | (x.xxx, x.xxx) | XXX | xxxxx | xxxxxx |

Source Program: xxxxxxx.sas

Table format is repeated for each reader. Entire table (all parts) is repeated for the PP population.

<sup>&</sup>lt;sup>a</sup> Change in ACR will be evaluated through the following components of the ACR Response Criteria: swollen joint count, tender joint count, patient assessment, physician assessment, pain scale, disability/functionality questionnaire, and acute phase reactant (ESR).

 $<sup>^{</sup> ext{b}}$  Kendall rank correlation between  $\Delta$ TUV at 24 weeks and the indicated measurement and time point.

<sup>&</sup>lt;sup>c</sup> Confidence limits calculated using Fisher's Z-transformation.

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 25. Frequency Counts of Localization in SPECT/CT Imaging in RA-2 Subjects
Navidea Biopharmaceuticals - Study No. NAV3-31

ITD Population (N=xxx)

#### Localized on SPECT/CT

| Reader | No | Yes | Total |
|--------|-------|-------|-------|
| xx | xxx | xxx | xxx |
| | XX.X% | XX.X% | |
| XX | xxx | xxx | XXX |
| | XX.X% | xx.x% | |
| XX | xxx | xxx | xxx |
| | xx.x% | XX.X% | |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format is repeated for the PP population.

Page x of y

Table 27. Number and Percentage of Subjects with TEAEs
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | | $\mathtt{Arm}^\mathtt{b}$ | | |
|---|---|---|---|---|
| Adverse Event Categorya: | HC | RA-2 | RA-3 | Overall |
| Total Number of TEAEs | xxx | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

b HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

# Table 28. Summary of TEAEs Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| | | Armb | | |
|---|---|---|---|---|
| | HC | RA-2 | RA-3 | Overall |
| Subjects With at Least One TEAE | xxx | xxx | xxx | xxx |
| Maximum TEAE Severity Grade | | | | |
| Mild | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Moderate | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Severe | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Tc 99m tilmanocept | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Study Procedure | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Subjects with at Least One TESAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

STATKING Clinical Services (DD-MMM-YYYY)

b HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Table 29. Number and Percentage of Subjects with TESAEs
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | | $\mathtt{Arm}^\mathtt{b}$ | | |
|---|---|---|---|---|
| Adverse Event Categorya: | HC | RA-2 | RA-3 | Overall |
| Total Number of TESAEs | xxx | xxx | xxx | xxx |
| Subjects with at Least One TESAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

b HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Table 30. Number and Percentage of Subjects With TEAEs by Severity Grade
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Part 1 of 4 - HCa

| | | Severity Grad | ie |
|---------------------------------|------------|---------------|------------|
| Adverse Event Categoryb: | Mild | Moderate | Severe |
| Total Number of TEAEs | xxx | xxx | XXX |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table format repeats for RA-2 and RA-3 (Parts 2 and 3) and overall (Part 4).

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b Adverse events coded with MedDRA Coding Dictionary Version XXX. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 31. Number and Percentage of Subjects With TEAEs by Level of Relationship to Tc 99m Tilmanocept

Navidea Biopharmaceuticals - Study No. NAV3-31

Safety Population (N=xxx)

Part 1 of 4 - HCa

Level of Relationship

| Adverse Event Category <sup>b</sup> : | Definitely<br>Not | Probably<br>Not | Possibly<br>Related | Probably<br>Related | Definitely<br>Related |
|---|---|---|---|---|---|
| Total Number of TEAEs | xxx | XXX | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format repeats for RA-2 and RA-3 (Parts 2 and 3) and overall (Part 4). Full Table (all parts) repeats for Table 32.

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 33. Serum Chemistry Clinical Laboratory Parameters Summary Statistics by Arm
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter(units) | Arma | Visit | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| xxxxxxxx (xxx) | HC | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 | RAW | | | | | | |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 8 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| xxxxxxxx (xxx) | HC | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 | RAW | | | | | | |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 8 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | xxxxxxxxx | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

Source Program: xxxxxxx.sas

Table format repeats for tables 34 and 35.

 $<sup>^{</sup>a}$  HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value). STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 36. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Part 1 of 7: Arm 1 HCa - Day 0

## Baseline Result/ Post-Injection Result

| Panel/Parameter (units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx (xxx)<br>xxxxxxx/<br>xxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

 $<sup>^{</sup>a}$  HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Table 36. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Part 2 of 7: Arm 2 RA-2a - Day 0

### Baseline Result/ Post-Injection Result

| Panel/Parameter (units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Table 36. Clinical Laboratory Parameters Shift Table by Arm Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

Part 3 of 7: Arm 2  $RA-2^a$  - Day 8

## Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

 $<sup>^{</sup>a}$  HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

Page x of y

Table 36. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Part 4 of 7: Arm 3 RA-3a - Day 0

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

Page x of y

Table 36. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Part 5 of 7: Arm RA-3a - Week 5

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| , | | ( 0) | ( 0) | | ( 0) | | ( 0) | ( 0) | ( 0) |
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx (xxx) | | | | | | | | | |
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx (xxx) | | | | | | | | | |
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx (xxx) | | | | | | | | | |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

Page x of y

Table 36. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Part 6 of 7: Arm 3 RA-3<sup>a</sup> - Week 12

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

Page x of y

Table 36. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Part 7 of 7: Arm 3 RA-3a - Week 24

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

<sup>&</sup>lt;sup>a</sup> HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

Page x of y

Table 39. ECG Parameters Summary Statistics by Arm Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| ECG | | | Data | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter(units) | ${\tt Arm^a}$ | Visit | Type <sup>b</sup> | Mean | Std Dev | n | Min | Max | Median |
| xxxxxxxxx (xxx) | HC | Day 0 Pre-Injection (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | Day 8 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 8 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Week 5 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Week 5 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Week 12 Pre-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | (Baseline) | | | | | | | |
| | | Week 12 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Week 24 Pre-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | (Baseline) | | | | | | | |
| | | Week 24 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | xxx | XXX | XXX | XXX | XXX | XXX |

<sup>&</sup>lt;sup>a</sup> HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

b RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value).

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas
Page x of y

Table 40. ECG Shift Table by Arm

Navidea Biopharmaceuticals - Study No. NAV3-31

Safety Population (N=xxx)

Baseline Result/
Post-Injection Result

| Arm | Visit | Abnormal/<br>Abnormal | Abnormal/<br>Normal | Normal/<br>Abnormal | Normal/<br>Normal |
|---|---|---|---|---|---|
| xxxx | xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| AAAA | XXXXX | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | XXXXX | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxx | xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | XXXXX | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxx | xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | xxxxx | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Table 41. Vital Signs Summary Statistics by Arm Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| Vital Sign | | | Data | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter (units) | ${\tt Arm^a}$ | Visit | $Type^b$ | Mean | Std Dev | n | Min | Max | Median |
| xxxxxxxxx (xxx) | HC | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-2 | Day 8 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 8 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Week 5 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Week 5 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Week 12 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Week 12 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA-3 | Week 24 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | xxx | XXX | XXX |
| | | Week 24 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

 $<sup>^{</sup>a}$  HC = healthy control, RA-2 = rheumatoid arthritis (stable treatment regimen), RA-3 = rheumatoid arthritis (candidate for changed treatment).

b RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value).

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 42. ACR Response Classification by Time Point Navidea Biopharmaceuticals - Study No. NAV3-31 ITD Population (N=xxx)

Arm 3 - RA-3ª Subjects Only

| | | Assessment | | |
|------------|------------|------------|------------|------------|
| Time Point | ACR-0 | ACR-20 | ACR-50 | ACR-70 |
| Week 5 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Week 12 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Week 24 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format Repeats for PP Population.

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Table 44. Concordance of  $\Delta TUV_{global[5w]}$  Bucketing and Week 12 Clinical Improvement Criteria Navidea Biopharmaceuticals - Study No. NAV3-31 ITD Population (N=xxx)

Arm 3 - RA-3ª Subjects Only

Part 1 of 6: ACR-20

| | Clinical | Assessment | | | |
|---|---|---|---|---|---|
| $\Delta ext{TUV}_{	ext{global}[5w]}$ Classification | Improved | Not<br>Improved | Total | Measure | Value <sup>b</sup> |
| Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Uncertainty Coefficient (C R) | xxxx (xxxxx) |
| Not Improved | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Uncertainty Coefficient (Symmetric) | xxxx (xxxxx) |
| Total | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | Positive Predictive Value<br>Confidence Limits | xxxx<br>(xxxx, xxxx) |
| | | | | Negative Predictive Value<br>Confidence Limits | xxxx<br>(xxxx, xxxx) |
| | | | | Overall Accuracy<br>Confidence Limits | xxxx<br>(xxxx, xxxx) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

This part repeats for Part 2 (ACR-50), Part 3 (ACR-70), Part 4 (CDAI), Part 5 (DAS28), and Part 6 (HAQ-DI) Full table format repeats for PP population (table 45) and for tables 46 - 65.

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

<sup>&</sup>lt;sup>b</sup> Values in parentheses are standard errors for the uncertainty coefficients, and p-values for positive predictive value and negative predictive value testing Ho:  $\pi$  = 0.6.

Page x of y

Table 66. ACPA Summary Statistics in Arm 3
Navidea Biopharmaceuticals - Study No. NAV3-31
ITD Population (N=xxx)

| Visit | Variable or Category <sup>a</sup> | Statistic | ITD Population (N=xxx) |
|---|---|---|---|
| Screening (Baseline) | Quantitative ACPA Level | Mean (Std Dev) | xxx (xxxx) |
| - | - | n | xxx |
| | | Median | xxx |
| | | (Min, Max) | (xxx, xxx) |
| | ACPA Level ≤ 70 | n (%) | xxx (xxx%) |
| | ACPA Level > 70 | n (%) | xxx (xxx%) |

## Table format repeats for PP population

<sup>&</sup>lt;sup>a</sup> Categories correspond to the ACPA bucketing levels used in the prediction of improvement algorithms. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Figure 1. Plot of  $\Delta TUV_{global}$  by Imaging Time Point and ACR-20 for Arm 3 Navidea Biopharmaceuticals - Study No. NAV3-31 ITD Population (N=xxx)



Responder status based on ACR-20 at each week. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Figure format repeats for Figures 2-5. Footnote text will be updated in each figure to correspond to the clinical assessment noted in the title (ACR-50, ACR-70, CDAI, or DAS28).

Page x of y

Data Listing 1. Subject Disposition Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31

| | Subject | | Date of<br>Completion or | |
|---|---|---|---|---|
| $\operatorname{Arm}^{\operatorname{a}}$ | No. | Disposition Status | Withdrawal | Withdrawal Reason |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxx | xxxx | ***** | xxxxxxxx | ***** |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 2. Inclusion/Exclusion Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31

| Arm <sup>a</sup> | Subject<br>No. | Did Subject<br>Meet All<br>Eligibility<br>Criteria? | Criterion Category | Criterion | Was a<br>Waiver<br>Granted? | Is Subject a<br>Screen<br>Failure? |
|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxx | xxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx | xxxx | xxxx |
| XXXXXX | XXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |
| XXXXXX | XXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |
| XXXXXX | XXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |

STATKING Clinical Services (DD-MMM-YYYY)

 $<sup>^{</sup>a}$  HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 3. Protocol Deviations Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31

| Arma | Subject<br>No. | Date of<br>Deviation | Deviation Description | Deviation Category<br>(Major/Minor) |
|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXX | ****************** | XXXXXXXXXX |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |
| xxxxxx | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 4. Demographics Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | Subject | Informed<br>Consent | Time from<br>Diagnosis<br>of RA | Date<br>of | Height | Weight | Age | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Arma | No. | Date/Time | (months) b | Birth | (inches) | (pounds) | (years) | Gender | Race | Ethnicity |
| XXXXXX | XXXX | XXXXXX | XXX | XXXXXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX |

a HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

<sup>&</sup>lt;sup>b</sup> Calculated as the difference between date of enrollment and date of RA diagnosis. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 5. Subjects Excluded from ITD Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
All Enrolled Subjects (N=xxx)

| Arma | Subject No. | Reason for Exclusion |
|--------|-------------|----------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 6. Subjects Excluded from PP Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
All Enrolled Subjects (N=xxx)

| Arma | Subject No. | Reason for Exclusion |
|--------|-------------|-------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 7. Subjects Excluded from Safety Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
All Enrolled Subjects (N=xxx)

| Arma | Subject No. | Reason for Exclusion |
|--------|-------------|-------------------------|
| · | | |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | xxxx | xxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 8. Medical History Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | | MedDRA System Organ Classb/ | | | |
|---|---|---|---|---|---|
| | Subject | MedDRA Preferred Term/ | | Resolution/Stop | o<br>O |
| Arma | No. | CRF Verbatim Term | Start Date | Date | Ongoing? |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

 $<sup>^{\</sup>rm b}$  Medical history terms coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 9. Prior and Concomitant Medications Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Drug Preferred Termb/

| | | | Verbatim/ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Subject | ATC Level 1 Text/ | | | Start | Stop | | |
| | $\mathtt{Arm}^\mathtt{a}$ | No. | ATC Level 4 Text | Indication | Frequency | Date | Date | Route | Ongoing? |
| , | | | | | | | | | |
| | XXXXXX | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b Medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 10. Prior and Concomitant RA Medications Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

Drug Preferred Termb/

| | | verbatim/ | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject | ATC Level 1 Text/ | | | Start | Stop | | |
| Arma | No. | ATC Level 4 Text | Indication | Frequency | Date | Date | Route | Ongoing? |
| XXXXXX | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| XXXXXX | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b Medications coded with WHO Coding Dictionary xxxxxxxx STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 11. Adverse Events Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | | | Start Date | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Start | and Time of | | MedDRA System Organ | | | | |
| | | Date and | Nearest | | Class <sup>b</sup> / | | Relation to | | |
| | | Time/ | Previous | | MedDRA Preferred | | Tc-99m | | |
| | Subject | End Date | tilmanocept | Treatment | Term/ | | tilmanocept/ | | |
| Arma | No. | and Time | Injection | Emergent? | CRF Verbatim Term | Severity | Procedure | Serious? | Outcome |
| XXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XXX | xxxxxxxxxxxxxx | XXXXXXXX | xxxxxxxx/ | XXX | XXXXXXXX |
| | | xxxxxxx/ | XXXXXXX | | xxxxxxxxxxxxxx | | XXXXXXX | | |
| | | XXXXXXX | | | xxxxxxxxxxxxxx | | | | |
| | | XXXXXXX | | | | | | | |
| XXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XXX | xxxxxxxxxxxxxxx | XXXXXXXX | xxxxxxxx/ | XXX | XXXXXXX |
| | | xxxxxxx/ | XXXXXXX | | xxxxxxxxxxxxxx | | XXXXXXX | | |
| | | XXXXXXX | | | xxxxxxxxxxxxxx | | | | |
| | | XXXXXXX | | | | | | | |

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 12. Subject Laboratory Profiles - Hematology Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | | | | | | | Norma | l Range | |
|---|---|---|---|---|---|---|---|---|---|
| _ | Arma | Subject<br>No. | Visit | Sample Date<br>and Time | Lab Parameter (Units) | Result | Lab Low | Lab High | Clin. Sig? |
| | XXXXXX | XXXX | XXXXXXX | xxxxxxxx / xx:xx | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |

 ${\tt STATKING~Clinical~Services~(DD-MMM-YYYY)}$ 

Source Program: xxxxxxx.sas

Table format is repeated for Serum Chemistry, Urinalysis, and Rheumatology Panel Listings (Listings 13, 14, 15).

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 16. Physical Exam Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | Subject | | Date | | | |
|---|---|---|---|---|---|---|
| ${\tt Arm^a}$ | No. | Visit | Conducted | Body System | Result | Abnormality |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | General Appearance | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Skin | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Eyes, Ears, Nose, Throat | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Head and Neck | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Lungs | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Heart | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Abdomen | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Lymph Nodes | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Musculoskeletal | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Nervous System | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Other: XXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 17. ACR/EULAR 2010 Classification Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

## ACR/EULAR 2010

| | Subject | | | Joint | | Acute-<br>Phase | Duration<br>of | |
|---|---|---|---|---|---|---|---|---|
| ${\tt Arm^a}$ | No. | Visit | Date | Involvement | Serology | Reactants | Symptoms | Total Score |
| xxxxxx | xxxx | xxxxxx | xxxxxx | xxx | xxx | xxx | xxx | xxx |
| xxxxxx | XXXX | xxxxxx | xxxxxx | xxx | xxx | xxx | xxx | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 18. ACR Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

ACR Components

| | | | | | | | <u>-</u> - | | | | • | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Patient's | Physician's | | Patient | Acute | | | |
| | | | | Tender | Swollen | Global | Global | Patient | Assessment | Phase | | | |
| | Subject | | | Joint | Joint | Disease | Disease | Assessment | Physical | Reactant | ACR- | ACR- | ACR- |
| Arma | No. | Visit | Date | Count | Count | Activity | Activity | of Pain | Function | Value | 20 | 50 | 70 |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 19. CDAI, DAS28, HAQ-DI, and WPI Scores Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| | | | | | CDAI | Component | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Patient's | Physician's | | | | | HAQ- | |
| | | | | Tender | Swollen | Global | Global | CDAI | | DAS28 | | DI | WPI |
| | Subject | | | Joint | Joint | Disease | Disease | Total | CDAI | Total | DAS28 | Total | Total |
| Arma | No. | Visit | Date | Score | Score | Activity | Activity | Score | Improved | Score | Improved | Score | Score |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXX | XXX | XXX | XXX | XXX | X | XX.X | X | XX.X | xx.x |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXX | XXX | XXX | xxx | XXX | X | XX.X | X | XX.X | XX.X |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 20. DAS28 by Joint Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

## DAS28 Joint Classification

| | Subject | | | | Result | Result |
|--------|---------|---------|---------|----------|--------------|-------------|
| Arma | No. | Visit | Date | Joint | (Right Body) | (Left Body) |
| • | | | | | | |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |
| | | | | XXXXXXXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 21. DAS28 by Subject Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| | | | | | | | DAS28 | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | • | | | Patient | Erythrocyte | |
| | | | | | Tender | Swollen | VAS | Sedimentation | |
| | | Subject | | | Joint | Joint | Global | Rate (ESR; | DAS28 |
| | Arma | No. | Visit | Date | Count | Count | (mm) | mm/hr) | Score |
| • | xxxxxx | xxxx | xxxxxx | xxxxxx | xxx | xxx | xxx | xxx | xxx |
| | xxxxxx | xxxx | xxxxxx | xxxxxx | xxx | xxx | xxx | XXX | xxx |

STATKING Clinical Services (DD-MMM-YYYY)

a HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 22. Vital Signs Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | Arm <sup>a</sup> | Subject<br>No. | Visit | Date | Time | Temp. | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Heart<br>Rate<br>(bpm) | Respirations<br>per Minute |
|---|---|---|---|---|---|---|---|---|---|---|
| ٠ | xxxxx | xxxx | xxxxxx | xxxxxx | xxxxx | xxx | xxx | XXX | xxx | xxx |
| | xxxxxx | xxxx | xxxxxx | xxxxxx | xxxxx<br>xxxxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx |
| | | | | | XXXXX | xxx | xxx | xxx<br>xxx | xxx | xxx<br>xxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 23. ECG Parameters Data Listing Navidea Biopharmaceuticals - Study No. NAV3-31 Safety Population (N=xxx)

| Arm <sup>a</sup> | Subject<br>No. | Visit | Date | Time | Heart Rate (bpm) | PR Interval (msec) | QRS<br>Interval<br>(msec) | QT Interval (msec) | QTcF<br>Interval<br>(msec) | Overall<br>Interpretation |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxx | xxxxx | xxxxxx | xxxxxx | xxxxxxx | xxxxxxx | xxxxxx | xxxx | xxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 24. Study Drug Administration Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| Arm <sup>a</sup> | Subject<br>No. | Date/<br>Time of<br>Injection | Anatomic<br>Location<br>of<br>Injection | Pre-Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Post-<br>Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Calculated Amount of Administered Radioactivity (mCi) | Calculated<br>Mass Dose<br>(µg) | Volume<br>Injected<br>(mL) | Lot<br>Number |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | xxx |
| xxxxxx | xxxx | xxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | xxx |
| | | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 25. Post-Injection Imaging Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| Arma | Subject<br>No. | Visit | Date of<br>Imaging | Start Time of Imaging | SPECT/CT Image<br>Finding | |
|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxx | xx:xx | xxx | _ |
| xxxxxx | xxxx | xxxxxxx | xxxxxx | xx:xx | XXX | |

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b SPECT/CT imaging performed only in study arm RA-2. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 26. SPECT/CT Reader Results Data Listing - Hands and Wrists
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| Arma | Subject<br>No. | Post-Injection<br>Imaging Time Point | Joint | SPECT/CT<br>Image Finding |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxx | xxxxxxxxxx | xxxx |
| xxxxxx | xxxx | xxxxxx | XXXXXXXXXXX<br>XXXXXXXXXXX | xxxx |

STATKING Clinical Services (DD-MMM-YYYY)

 $<sup>^{</sup>a}$  HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

Page x of y

Data Listing 27. TUV Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

TUV Classification of Improvement

| Arm <sup>a</sup> | Subject No. | Algorithms<br>Predicting<br>Improvement <sup>b</sup> | Algorithms<br>Predicting No<br>Improvement <sup>b</sup> | Reader<br>No. | Visit | Date/Time | Region of<br>Interest <sup>c</sup> | TUV |
|---|---|---|---|---|---|---|---|---|
| | VVVV | v v v | v v v | | .,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | WWW.WW | |
| XXXXXX | XXXX | X, X, X | x, x, x, x | XXX | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| | | | | XXX | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| | | | | XXX | xxxxxxx | XXXXXX | xxxxxx | xxxxx |
| | | | | XXX | XXXXXXX | XXXXXX | XXXXXX | XXXXX |
| XXXXXX | XXXX | X | X, $X$ , $X$ , $X$ , $X$ , $X$ | XXX | XXXXXXX | XXXXXX | XXXXXX | XXXXX |

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b 1 = Change in Global TUV(5w) Bucketing, 2 = Change in Global TUV(5w), 3 = Change in Global TUV(5w) Bucketing with ACPA Bucketing, 4 = Change in Global TUV(12w) Bucketing, 5 = Change in Global TUV(12w), 6 = Change in Global TUV(12w) Bucketing with ACPA Bucketing, 7 = ACPA Bucketing Alone.

 $<sup>^{\</sup>circ}$  Region of Interest is joint for all arms, and joint or Global for the RA-2 and RA-3 arms. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 28. ACR Response Criteria Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-31
Safety Population (N=xxx)

| | Subject | | ACR Response | Number of<br>Tender | Number of<br>Swollen | Patient<br>Global | Physician<br>Global | | VAS Pain | |
|---|---|---|---|---|---|---|---|---|---|---|
| Arma | No. | Visit | Assessment <sup>b</sup> | Joints | Joints | Assessment | Assessment | HAQ Total | Score | ESR |
| XXXXXX | XXXX | XXXXXXX | xxxxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXXX | XXXXXXX | xxxxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC = Healthy Control, RA-2 = Rheumatoid Arthritis (stable treatment regimen), RA-3 = Rheumatoid Arthritis (candidate for changed treatment).

b Response assessment will be blank for baseline measurements.